CLINICAL TRIAL: NCT03758313
Title: Non-Invasive Monitoring of Partial Pressure of Carbon Dioxide in Mechanically Ventilated Preterm Infants
Status: Completed | Type: Observational
Sponsor: Tobias Werther (Other)
Responsible Party: Sponsor-Investigator, Tobias Werther, Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: 1173/2018
Record Dates: First submitted 2018-11-26; First posted 2018-11-29 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Preterm Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CO2 measurements — Distal etCO2, tcCO2 and paCO2 values will be recorded simultaneously in ventilated preterm infants. We will measure etCO2 in a distal position using a double lumen tube connected to an external side-stream capnometer.

SUMMARY:
In mechanically ventilated preterm infants, the ability to monitor carbon dioxide partial pressure (pCO2) values is indispensable. The gold standard for pCO2 measurement is from an arterial blood sample (paCO2). This has two drawbacks: firstly, it requires an arterial line and, secondly, it does not provide the clinicians with a continuous measurement. At present, two alternative pCO2 monitoring systems are available in the field of neonatal intensive care medicine: end-tidal CO2 (etCO2) capnography and transcutaneous CO2 (tcCO2) measurements. Both methods have disadvantages including potential technical errors as well as pathologies that may reduce reliability as a surrogate for blood gas analysis (BGA). In particular, conventional side-stream etCO2 capnography underestimates pCO2 in presence of a tube leakage, which is a common occurrence in ventilated preterm infants where only tubes without cuff are used. Distal etCO2 (detCO2) by means of a double lumen endo-tracheal tube may solve the problem of unreliable etCO2 values in the presence of tube leakage.

The aim of this study is to compare the agreement, precision and repeatability of the distal etCO2-measurement technique described by Kugelman et al. with respect to paCO2 and tcCO2 in mechanically ventilated preterm infants. Since ventilation strategies and pCO2 limits may vary among different centers, this study helps to determine which non-invasive CO2 monitoring system (detCO2 or tcO2) is more suitable in terms of applicability and reliability in preterm infants at our neonatal intensive care units.

DETAILED DESCRIPTION:
Background: In mechanically ventilated preterm infants, the ability to monitor carbon dioxide partial pressure (pCO2) values is indispensable. The gold standard for pCO2 measurement is from an arterial blood sample (paCO2). This has two drawbacks: firstly, it requires an arterial line and, secondly, it does not provide the clinicians with a continuous measurement. At present, two alternative pCO2 monitoring systems are available in the field of neonatal intensive care medicine: end-tidal CO2 (etCO2) capnography and transcutaneous CO2 (tcCO2) measurements. Both methods have disadvantages including potential technical errors as well as pathologies that may reduce reliability as a surrogate for blood gas analysis (BGA). In particular, conventional side-stream etCO2 capnography underestimates pCO2 in presence of a tube leakage, which is a common occurrence in ventilated preterm infants where only tubes without cuff are used. Distal etCO2 (detCO2) by means of a double lumen endo-tracheal tube may solve the problem of unreliable etCO2 values in the presence of tube leakage.

Several studies compared etCO2 and tcCO2 to paCO2, simultaneously. A comparison study of etCO2 and tcCO2 in a cohort of critically ill children did not reveal significant differences in the absence of severe pulmonary parenchymal disease. Tobias et al compared etCO2 and tcCO2 in a cohort of pediatric intensive care patients with respiratory failure and found tcCO2 measurements to be more accurate. In a cohort of ventilated newborns, tcCO2 monitoring was generally more precise than etCO2 during neonatal transport to monitor ventilation. In a more recent study restricted to a cohort of postsurgical neonates without lung disease, etCO2 underestimated paCO2 more than tcCO2 but provided greater precision over paCO2, however it was less accurate at smaller tidal volumes. These studies have in common that the adapter of the pCO2 analyzer was attached in-line and proximal to the endotracheal tube.

Aim of the study: The aim of this study is to compare the agreement, precision and repeatability of the distal etCO2-measurement technique described by Kugelman et al. with respect to paCO2 and tcCO2 in mechanically ventilated preterm infants. Since ventilation strategies and pCO2 limits may vary among different centers, this study helps to determine which non-invasive CO2 monitoring system (detCO2 or tcO2) is more suitable in terms of applicability and reliability in preterm infants at our neonatal intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with a current body weight between 1000 g and 3000 g who require intubation.
* Signed informed consent from parents or legal guardians.
* Expected to provide at least three measurements of paCO2 and detCO2.

Exclusion Criteria:

* Infants with known congenital anomalies of the heart and/or lung.
* Need for high frequency oscillation.
* Parents or legal guardians deny informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mechanically Ventilated Preterm Infants
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Carbon Dioxide in Mechanically Ventilated Preterm Infants | 48 hours
  partial pressure of carbon dioxide

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Werther, PhD, Principal Investigator — Medical University Vienna
Locations (1):
- Department of Pediatrics, Division of Neonatology, Pediatric Intensive Care and Neuropediatrics, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Morley CJ, Davis PG, Doyle LW, Brion LP, Hascoet JM, Carlin JB; COIN Trial Investigators. Nasal CPAP or intubation at birth for very preterm infants. N Engl J Med. 2008 Feb 14;358(7):700-8. doi: 10.1056/NEJMoa072788. PMID 18272893
- [Background] Giannakopoulou C, Korakaki E, Manoura A, Bikouvarakis S, Papageorgiou M, Gourgiotis D, Hatzidaki E. Significance of hypocarbia in the development of periventricular leukomalacia in preterm infants. Pediatr Int. 2004 Jun;46(3):268-73. doi: 10.1111/j.1442-200x.2004.01886.x. PMID 15151541
- [Background] Erickson SJ, Grauaug A, Gurrin L, Swaminathan M. Hypocarbia in the ventilated preterm infant and its effect on intraventricular haemorrhage and bronchopulmonary dysplasia. J Paediatr Child Health. 2002 Dec;38(6):560-2. doi: 10.1046/j.1440-1754.2002.00041.x. PMID 12410866
- [Background] Tobias JD. Transcutaneous carbon dioxide monitoring in infants and children. Paediatr Anaesth. 2009 May;19(5):434-44. doi: 10.1111/j.1460-9592.2009.02930.x. Epub 2009 Feb 19. PMID 19236597
- [Background] Aliwalas LL, Noble L, Nesbitt K, Fallah S, Shah V, Shah PS. Agreement of carbon dioxide levels measured by arterial, transcutaneous and end tidal methods in preterm infants < or = 28 weeks gestation. J Perinatol. 2005 Jan;25(1):26-9. doi: 10.1038/sj.jp.7211202. PMID 15496874
- [Background] Molloy EJ, Deakins K. Are carbon dioxide detectors useful in neonates? Arch Dis Child Fetal Neonatal Ed. 2006 Jul;91(4):F295-8. doi: 10.1136/adc.2005.082008. PMID 16790735
- [Background] McDonald MJ, Montgomery VL, Cerrito PB, Parrish CJ, Boland KA, Sullivan JE. Comparison of end-tidal CO2 and Paco2 in children receiving mechanical ventilation. Pediatr Crit Care Med. 2002 Jul;3(3):244-249. doi: 10.1097/00130478-200207000-00008. PMID 12780964
- [Background] Schmalisch G. Current methodological and technical limitations of time and volumetric capnography in newborns. Biomed Eng Online. 2016 Aug 30;15(1):104. doi: 10.1186/s12938-016-0228-4. PMID 27576441
- [Background] Anderson CT, Breen PH. Carbon dioxide kinetics and capnography during critical care. Crit Care. 2000;4(4):207-15. doi: 10.1186/cc696. Epub 2000 Jul 12. PMID 11094503
- [Background] Wu CH, Chou HC, Hsieh WS, Chen WK, Huang PY, Tsao PN. Good estimation of arterial carbon dioxide by end-tidal carbon dioxide monitoring in the neonatal intensive care unit. Pediatr Pulmonol. 2003 Apr;35(4):292-5. doi: 10.1002/ppul.10260. PMID 12629627
- [Background] Amuchou Singh S, Singhal N. Dose end-tidal carbon dioxide measurement correlate with arterial carbon dioxide in extremely low birth weight infants in the first week of life? Indian Pediatr. 2006 Jan;43(1):20-5. PMID 16465002
- [Background] Dargaville PA, Tingay DG. Lung protective ventilation in extremely preterm infants. J Paediatr Child Health. 2012 Sep;48(9):740-6. doi: 10.1111/j.1440-1754.2012.02532.x. PMID 22970667
- [Background] Keszler M, Nassabeh-Montazami S, Abubakar K. Evolution of tidal volume requirement during the first 3 weeks of life in infants <800 g ventilated with Volume Guarantee. Arch Dis Child Fetal Neonatal Ed. 2009 Jul;94(4):F279-82. doi: 10.1136/adc.2008.147157. Epub 2008 Dec 5. PMID 19060010
- [Background] Nassabeh-Montazami S, Abubakar KM, Keszler M. The impact of instrumental dead-space in volume-targeted ventilation of the extremely low birth weight (ELBW) infant. Pediatr Pulmonol. 2009 Feb;44(2):128-33. doi: 10.1002/ppul.20954. PMID 19061234
- [Background] Hagerty JJ, Kleinman ME, Zurakowski D, Lyons AC, Krauss B. Accuracy of a new low-flow sidestream capnography technology in newborns: a pilot study. J Perinatol. 2002 Apr-May;22(3):219-25. doi: 10.1038/sj.jp.7210672. PMID 11948385
- [Background] Nangia S, Saili A, Dutta AK. End tidal carbon dioxide monitoring--its reliability in neonates. Indian J Pediatr. 1997 May-Jun;64(3):389-94. doi: 10.1007/BF02845211. PMID 10771861
- [Background] Singh BS, Gilbert U, Singh S, Govindaswami B. Sidestream microstream end tidal carbon dioxide measurements and blood gas correlations in neonatal intensive care unit. Pediatr Pulmonol. 2013 Mar;48(3):250-6. doi: 10.1002/ppul.22593. Epub 2012 May 15. PMID 22589000
- [Background] Mahmoud RA, Proquitte H, Fawzy N, Buhrer C, Schmalisch G. Tracheal tube airleak in clinical practice and impact on tidal volume measurement in ventilated neonates. Pediatr Crit Care Med. 2011 Mar;12(2):197-202. doi: 10.1097/PCC.0b013e3181e89834. PMID 20581731
- [Background] Schmalisch G, Al-Gaaf S, Proquitte H, Roehr CC. Effect of endotracheal tube leak on capnographic measurements in a ventilated neonatal lung model. Physiol Meas. 2012 Oct;33(10):1631-41. doi: 10.1088/0967-3334/33/10/1631. Epub 2012 Sep 18. PMID 22986303
- [Background] Proquitte H, Krause S, Rudiger M, Wauer RR, Schmalisch G. Current limitations of volumetric capnography in surfactant-depleted small lungs. Pediatr Crit Care Med. 2004 Jan;5(1):75-80. doi: 10.1097/01.PCC.0000102384.60676.E5. PMID 14697113
- [Background] Kugelman A, Golan A, Riskin A, Shoris I, Ronen M, Qumqam N, Bader D, Bromiker R. Impact of Continuous Capnography in Ventilated Neonates: A Randomized, Multicenter Study. J Pediatr. 2016 Jan;168:56-61.e2. doi: 10.1016/j.jpeds.2015.09.051. Epub 2015 Oct 17. PMID 26490126
- [Background] Kugelman A, Zeiger-Aginsky D, Bader D, Shoris I, Riskin A. A novel method of distal end-tidal CO2 capnography in intubated infants: comparison with arterial CO2 and with proximal mainstream end-tidal CO2. Pediatrics. 2008 Dec;122(6):e1219-24. doi: 10.1542/peds.2008-1300. Epub 2008 Nov 24. PMID 19029196
- [Background] Cassady G. Transcutaneous monitoring in the newborn infant. J Pediatr. 1983 Dec;103(6):837-48. doi: 10.1016/s0022-3476(83)80698-2. No abstract available. PMID 6417293
- [Background] Rennie JM. Transcutaneous carbon dioxide monitoring. Arch Dis Child. 1990 Apr;65(4 Spec No):345-6. doi: 10.1136/adc.65.4_spec_no.345. No abstract available. PMID 2110802
- [Background] Bendjelid K, Schutz N, Stotz M, Gerard I, Suter PM, Romand JA. Transcutaneous PCO2 monitoring in critically ill adults: clinical evaluation of a new sensor. Crit Care Med. 2005 Oct;33(10):2203-6. doi: 10.1097/01.ccm.0000181734.26070.26. PMID 16215371
- [Background] Dullenkopf A, Bernardo SD, Berger F, Fasnacht M, Gerber AC, Weiss M. Evaluation of a new combined SpO2/PtcCO2 sensor in anaesthetized paediatric patients. Paediatr Anaesth. 2003 Nov;13(9):777-84. doi: 10.1046/j.1460-9592.2003.01146.x. PMID 14617118
- [Background] Sorensen LC, Brage-Andersen L, Greisen G. Effects of the transcutaneous electrode temperature on the accuracy of transcutaneous carbon dioxide tension. Scand J Clin Lab Invest. 2011 Nov;71(7):548-52. doi: 10.3109/00365513.2011.590601. Epub 2011 Jul 6. PMID 21732731
- [Background] Eberhard P. The design, use, and results of transcutaneous carbon dioxide analysis: current and future directions. Anesth Analg. 2007 Dec;105(6 Suppl):S48-S52. doi: 10.1213/01.ane.0000278642.16117.f8. PMID 18048898
- [Background] Hirata K, Nishihara M, Oshima Y, Hirano S, Kitajima H. Application of transcutaneous carbon dioxide tension monitoring with low electrode temperatures in premature infants in the early postnatal period. Am J Perinatol. 2014 May;31(5):435-40. doi: 10.1055/s-0033-1352485. Epub 2013 Aug 5. PMID 23918520
- [Background] Aly S, El-Dib M, Mohamed M, Aly H. Transcutaneous Carbon Dioxide Monitoring with Reduced-Temperature Probes in Very Low Birth Weight Infants. Am J Perinatol. 2017 Apr;34(5):480-485. doi: 10.1055/s-0036-1593352. Epub 2016 Sep 27. PMID 27673754
- [Background] Karlsson V, Sporre B, Agren J. Transcutaneous PCO2 Monitoring in Newborn Infants During General Anesthesia Is Technically Feasible. Anesth Analg. 2016 Oct;123(4):1004-7. doi: 10.1213/ANE.0000000000001462. PMID 27464976
- [Background] Restrepo RD, Hirst KR, Wittnebel L, Wettstein R. AARC clinical practice guideline: transcutaneous monitoring of carbon dioxide and oxygen: 2012. Respir Care. 2012 Nov;57(11):1955-62. doi: 10.4187/respcare.02011. PMID 23107301
- [Background] Sivan Y, Eldadah MK, Cheah TE, Newth CJ. Estimation of arterial carbon dioxide by end-tidal and transcutaneous PCO2 measurements in ventilated children. Pediatr Pulmonol. 1992 Mar;12(3):153-7. doi: 10.1002/ppul.1950120305. PMID 1641271
- [Background] Tobias JD, Meyer DJ. Noninvasive monitoring of carbon dioxide during respiratory failure in toddlers and infants: end-tidal versus transcutaneous carbon dioxide. Anesth Analg. 1997 Jul;85(1):55-8. doi: 10.1097/00000539-199707000-00010. PMID 9212122
- [Background] Tingay DG, Stewart MJ, Morley CJ. Monitoring of end tidal carbon dioxide and transcutaneous carbon dioxide during neonatal transport. Arch Dis Child Fetal Neonatal Ed. 2005 Nov;90(6):F523-6. doi: 10.1136/adc.2004.064717. Epub 2005 Apr 29. PMID 15863489
- [Background] Tingay DG, Mun KS, Perkins EJ. End tidal carbon dioxide is as reliable as transcutaneous monitoring in ventilated postsurgical neonates. Arch Dis Child Fetal Neonatal Ed. 2013 Mar;98(2):F161-4. doi: 10.1136/fetalneonatal-2011-301606. Epub 2012 Aug 11. PMID 22887048
- [Background] van Kaam AH, De Jaegere AP, Rimensberger PC; Neovent Study Group. Incidence of hypo- and hyper-capnia in a cross-sectional European cohort of ventilated newborn infants. Arch Dis Child Fetal Neonatal Ed. 2013 Jul;98(4):F323-6. doi: 10.1136/archdischild-2012-302649. Epub 2012 Dec 14. PMID 23241364
- [Background] Donner A, Eliasziw M. Sample size requirements for reliability studies. Stat Med. 1987 Jun;6(4):441-8. doi: 10.1002/sim.4780060404. PMID 3629046
- [Background] Muller R, Buttner P. A critical discussion of intraclass correlation coefficients. Stat Med. 1994 Dec 15-30;13(23-24):2465-76. doi: 10.1002/sim.4780132310. PMID 7701147
- [Background] Walter SD, Eliasziw M, Donner A. Sample size and optimal designs for reliability studies. Stat Med. 1998 Jan 15;17(1):101-10. doi: 10.1002/(sici)1097-0258(19980115)17:13.0.co;2-e. PMID 9463853
- [Background] McSwain SD, Hamel DS, Smith PB, Gentile MA, Srinivasan S, Meliones JN, Cheifetz IM. End-tidal and arterial carbon dioxide measurements correlate across all levels of physiologic dead space. Respir Care. 2010 Mar;55(3):288-93. PMID 20196877
- [Background] Siobal MS. Monitoring Exhaled Carbon Dioxide. Respir Care. 2016 Oct;61(10):1397-416. doi: 10.4187/respcare.04919. Epub 2016 Sep 6. PMID 27601718
- [Background] Fayoux P, Devisme L, Merrot O, Marciniak B. Determination of endotracheal tube size in a perinatal population: an anatomical and experimental study. Anesthesiology. 2006 May;104(5):954-60. doi: 10.1097/00000542-200605000-00011. PMID 16645447
- [Background] Yildizdas D, Yapicioglu H, Yilmaz HL, Sertdemir Y. Correlation of simultaneously obtained capillary, venous, and arterial blood gases of patients in a paediatric intensive care unit. Arch Dis Child. 2004 Feb;89(2):176-80. doi: 10.1136/adc.2002.016261. PMID 14736638
- [Background] Zavorsky GS, Cao J, Mayo NE, Gabbay R, Murias JM. Arterial versus capillary blood gases: a meta-analysis. Respir Physiol Neurobiol. 2007 Mar 15;155(3):268-79. doi: 10.1016/j.resp.2006.07.002. Epub 2006 Aug 17. PMID 16919507
- [Background] Bland JM, Altman DG. Agreement between methods of measurement with multiple observations per individual. J Biopharm Stat. 2007;17(4):571-82. doi: 10.1080/10543400701329422. PMID 17613642
- [Derived] Werther T, Aichhorn L, Stellberg S, Cardona FS, Klebermass-Schrehof K, Berger A, Schmolzer GM, Wagner M. Monitoring of carbon dioxide in ventilated neonates: a prospective observational study. Arch Dis Child Fetal Neonatal Ed. 2022 May;107(3):293-298. doi: 10.1136/archdischild-2021-322138. Epub 2021 Aug 3. PMID 34344835